CLINICAL TRIAL: NCT05511519
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Zunsemetinib vs Placebo in Patients With Moderate-to-Severe Active Psoriatic Arthritis
Brief Title: Study of ATI-450 vs Placebo in Patients With Moderate to Severe Psoriatic Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-450-PsA-201
Record Dates: First submitted 2022-07-29; First posted 2022-08-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Psoriatic Arthritis
Keywords: Arthritis; Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded placebo drug is packaged to match the active study drug and will be stored under the same conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-450 (Experimental): ATI-450 50mg oral tablet BID
  Interventions: Drug: ATI-450
- Placebo (Placebo Comparator): Placebo oral tablet BID
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ATI-450 — Oral, small molecule MK2 inhibitor
  Other Names: CDD-450
  Arms: ATI-450
Drug: Placebo Oral Tablet — Placebo tablet manufactured to match ATI-450 in appearance
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to investigate the efficacy, safety, tolerability, PK, and PD of ATI-450 versus placebo in patients with moderate to severe psoriatic arthritis.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled study to investigate the efficacy, safety, tolerability, PK, and PD of ATI-450 versus placebo in patients with moderate to severe psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PsA with symptom onset at least 6 months before the Screening Visit and fulfilment of the Classification Criteria for PsA.
* Patient has moderate-to-severe PsA at Screening and Randomization Visits defined as

  * ≥3 tender joints (based on 68 joint counts) and
  * ≥3 swollen joints (based on 66 joint counts).
* Diagnosis of active plaque psoriasis or documented history of plaque psoriasis.

Exclusion Criteria:

* Any arthritis with onset before age 17 years, or current diagnosis of inflammatory joint disease other than PsA, or other immunological disease (including, but not limited to rheumatoid arthritis, gout, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, systemic lupus erythematosus).
* Patient has an uncontrolled non-immunoinflammatory disease that may place the patient at increased risk during the study or impact the interpretation of results, eg, cirrhosis, previous malignancy, previous venous thromboembolism.
* Any clinically significant laboratory abnormality that would affect interpretation of study data or safety of the patient's participation in the study, per judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving ACR20 at Week 12 | Baseline to Week 12

SECONDARY OUTCOMES:
Proportion of patients with ACR 50/70 at Week 12 | Baseline to Week 12
Proportion of patients with ACR 20/50/70 response at weeks 2, 4, 6, 8 | Baseline to Week 12
Change from baseline in tender joint count 68 at weeks 1, 2, 4, 6, 8, 12 | Baseline to Week 12
Change from baseline in swollen joint count 66 at weeks 1, 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Health Assessment Questionnaire - Disability Index at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in patient's global assessment of disease activity at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in physician's global assessment of disease activity at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Patients Pain VAS assessment at Weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in high sensitivity C-reactive protein (hs-CRP) at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Leeds Enthesitis Index over 12 weeks | Baseline to Week 12
Change from baseline in Leeds Dactylitis Index over 12 weeks | Baseline to Week 12
Proportion of patients achieving at least a 30% reduction and at least 1 unit reduction from Baseline in the numerical rating scale (NRS30) in Patient's Daily Assessment of Skin Pain at Weeks 2, 4, 8, 12 among patients with Baseline NRS ≥3 | Baseline to Week 12
Proportion of patients achieving a sIGA of Psoriasis of 0 or 1 and at least a 2-point improvement from baseline among those with a baseline investigator's global assessment of at least 3 over 12 weeks | Baseline to Week 12
Proportion of patients achieving MDA at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in DAS28CRP at Weeks 2, 4, 8, 12 | Baseline to Week 12
Psoriasis Area Severity Index (PASI) 50/75/90 response (for patients with ≥3% body surface area psoriasis at baseline) at Week 12 | Baseline to Week 12
Mean change from baseline in PASI score at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Short-Form-36 Physical Component Summary at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Functional Assessment of Chronic Illness Therapy-Fatigue Questionnaire at weeks 2, 4, 8, 12 | Baseline to Week 12
Change from baseline in Self-Assessment of Psoriasis Symptoms Questionnaire at weeks 2, 4, 8, 12 | Baseline to Week 12
Type and frequency of adverse events | Baseline to Week 12
Type and frequency of serious adverse events | Baseline to Week 12
Zunsemetinib trough concentration ng/mL | Baseline to Week 12
CDD-2164 metabolite trough concentration ng/mL | Baseline to Week 12
Zunsemetinib peak concentration (Cmax) ng/mL | Baseline to Week 12
CDD-2164 metabolite peak concentration (Cmax) ng/mL | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (20):
- United States (8):
  - Aclaris Investigational Site, Miami Lakes, Florida
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Clinical Operations, Freehold, New Jersey
  - Aclaris Clinical Operations, Charlotte, North Carolina
  - Aclaris Investigational Site, Perrysburg, Ohio
  - Aclaris Investigational Site, Duncansville, Pennsylvania
  - Aclaris Investigational Site, Memphis, Tennessee
  - Aclaris Investigational Site, Mesquite, Texas
- Poland (12):
  - Aclaris Investigational Site, Bialystok
  - Aclaris Investigational Site, Bydgoszcz
  - Aclaris Investigational Site, Częstochowa
  - Aclaris Investigational Site, Katowice
  - Aclaris Investigational Site, Krakow
  - Aclaris Investigational Site, Olsztyn
  - Aclaris Investigational Site, Poznan
  - Aclaris Investigational Site, Stalowa Wola
  - Aclaris Investigational Site, Szczecin
  - Aclaris Investigational Site, Torun
  - Aclaris Investigational Site, Warsaw
  - Aclaris Investigational Site, Wroclaw